CLINICAL TRIAL: NCT00990366
Title: Treatment of Biliary Obstruction Using Biliary Stent With or Without Antireflux Valve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis results, study terminated 5/2010
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hanna Vihervaara, Ph.D., Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58/180/2009
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Biliary Obstruction; Cholangitis
Keywords: antireflux valve; biliary obstruction; cholangitis; biliary stent
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- biliary stent without an antireflux valve (Active Comparator): patients with biliary obstruction who need a biliary stent, selected for the stent without an antireflux valve arm
  Interventions: Device: Cook´s biliary stent with an antireflux stent, normal biliary stent
- biliary stent with an antireflux valve (Active Comparator): patients with biliary obstruction, who need a biliary stent, selected for the stent with an antireflux valve arm
  Interventions: Device: Cook´s biliary stent with an antireflux stent, normal biliary stent

INTERVENTIONS:
Device: Cook´s biliary stent with an antireflux stent, normal biliary stent — arms are assigned randomly by closed envelope method

SUMMARY:
Biliary obstruction can be relieved by biliary stent. Ascending infection of biliary passage (cholangitis) causes hospitalization and obstruction of stents. Reflux of intestinal fluids through a stent is thought to be one of the causes of cholangitis. Stents with antireflux valves are designed to reduce the reflux from the bowel. The purpose of the study is to investigate prospectively whether it is possible to reduce the amount of infection and thus obstruction of biliary stent by using a stent with an antireflux valve compared to a normal stent without an antireflux valve.

ELIGIBILITY:
Inclusion Criteria:

* age 18-89
* biliary obstruction in the lower two thirds of the choledochus

Exclusion Criteria:

* allergy to contrast media
* future pancreaticoduodenectomy
* refusal from the study
* previous stent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
patency of a biliary stent | one year

SECONDARY OUTCOMES:
Cholangitis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Salminen, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland